CLINICAL TRIAL: NCT02289196
Title: A Multicenter, Open Label, Uncontrolled Phase I Trial to Compare Safety, Tolerability and Immunogenicity of Vx-006 Vaccine at 0.5mg, 1mg, 5mg and 10mg Doses in Human Leukocyte Antigen-A02 (HLA-A02) Positive Patients With Solid Tumours
Brief Title: Safety Study of Vx006 Vaccine in Solid Tumor Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vaxon Biotech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Vx-006-101
Record Dates: First submitted 2014-10-30; First posted 2014-11-13 (Estimated); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Solid Tumor
Keywords: Vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Vx-006: 0,5mg (Experimental): Six injections of Vx-006 at 0,5 mg + Montanide ISA51™ will be administrated every 3 weeks
  Interventions: Drug: Vx-006: 0,5mg
- Vx-006: 1mg (Experimental): Six injections of Vx-006 at 1 mg + Montanide ISA51™ will be administrated every 3 weeks
  Interventions: Drug: Vx-006: 1mg
- Vx-006: 5mg (Experimental): Six injections of Vx-006 at 5 mg + Montanide ISA51™ will be administrated every 3 weeks
  Interventions: Drug: Vx-006: 5mg
- Vx-006: 10mg (Experimental): Six injections of Vx-006 at 10 mg + Montanide ISA51™ will be administrated every 3 weeks
  Interventions: Drug: Vx-006: 10mg

INTERVENTIONS:
Drug: Vx-006: 0,5mg
  Arms: Vx-006: 0,5mg
Drug: Vx-006: 1mg
  Arms: Vx-006: 1mg
Drug: Vx-006: 5mg
  Arms: Vx-006: 5mg
Drug: Vx-006: 10mg
  Arms: Vx-006: 10mg

SUMMARY:
Patients with histologically proven malignancy with documented disease control (objective response or stable disease) or Not Evaluable Disease (NED) expectancy > 6 months; only HLA-A*02 positive patients.

The primary objective of the trial is to compare safety and tolerability of four different doses of Vx-006. The secondary objective is to compare immunogenicity of four different doses of the Vx-006.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female > or = 18 years of age;
2. Histologically proven malignancy;
3. Documented HLA-A*02 positivity, as determined by a central laboratory;
4. Disease control (Complete Response (CR), Partial Response (PR), or Stable Disease (SD)) according to Response Evaluation Criteria In Solid Tumors (RECIST 1.1) criteria or NED in the case of patients who received adjuvant chemotherapy
5. Patient with disease control or NED expectancy > or = 6 months according to investigator opinion;
6. ECOG performance status 0, 1;
7. Patients must have adequate renal and hepatic function as assessed by standard laboratory criteria;
8. Patients must have adequate haematological function:

   * Platelet count > or = 100 x 109/L;
   * White Blood Cell (WBC) count > or = 2.5 x 109/L;
   * Haemoglobin > or = 90g /L;
9. Female patients must be of non-child-bearing potential (i.e., women with functioning ovaries who have a documented tubal ligation or hysterectomy, ovariectomy or women who are post-menopausal). Women of child-bearing potential must have a negative urine pregnancy test at baseline and agree to practice adequate contraception for 30 days prior to administration of investigational product, throughout the study treatment period and 30 days after completion of injections;
10. In the investigator's opinion, the patient is capable and willing to comply with the requirements of the study;
11. Willing and able to sign a written informed consent.

Exclusion Criteria:

1. Prior treatment with cancer vaccines;
2. Treatment with immunotherapy (e.g., interferons, interleukins, Tumor Necrosis Factor (TNF), or biological response modifiers, such as Granulocyte-Macrophage Colony Stimulating Factor (GM-CSF) etc) within four weeks prior to the first vaccination;
3. Treatment with immunosuppressive agents (including corticosteroids) within 2 weeks prior to the first vaccination;
4. Treatment with any investigational drugs, within 4 weeks prior to the first vaccination;
5. Autoimmune or immunodeficiency disease that in the opinion of the investigator may compromise the safety of the patient in the study;
6. Any pre-existing medical condition requiring concomitant systemic corticosteroid or immunosuppressive therapy. The use of inhaled corticosteroids for Chronic Obstructive Pulmonary Disease (COPD) or topical steroids is allowed;
7. Known hepatitis B and/or C infection documented in patient files, testing not required;
8. Known HIV-positivity, testing not required;
9. Clinically significant hepatic dysfunction (Alanine amino transferase (ALT)>2.5 times normal upper limits [ULN], Aspartate Amino Transferase (AST)>2.5 times Upper Limit of Normal (ULN), bilirubin>1.5 times ULN);
10. Clinically significant renal dysfunction (serum creatinine>1.5 time ULN);
11. Uncontrolled congestive heart failure or hypertension, unstable heart disease (coronary artery disease with unstable angina or myocardial infarction within 6 months before enrolment) or uncontrolled ventricular arrhythmias at the time of enrolment in the study (atrial fibrillation or flutter is acceptable);
12. Splenectomy or splenic irradiation;
13. Any infectious condition that, in the opinion of the investigator, could compromise the patient's ability to develop an immune response;
14. Pregnant or lactating females (female patients of child-bearing potential will undertake pregnancy testing at screening and during study completion/withdrawal visits);
15. Alcohol or drug dependence;
16. Requirement of concurrent treatment with prohibited medication (investigational product, other anti-cancer treatments including chemotherapy, non-palliative radiotherapy, biological agents and immunomodulating agents, systemic immunosuppressive agents, including systemic corticosteroids);
17. The investigator considers the patient unfit for the study as a result of the medical interview, physical examination, or screening investigations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-03; Primary Completion 2014-10 (Actual); Study Completion 2017-05 (Actual)

PRIMARY OUTCOMES:
Adverse event number by treatment group as a measure of safety and tolerability | 18 Weeks
  The following parameters of safety and tolerability will be assessed:
  * Physical examination and vital signs (blood pressure, pulse rate, body temperature, weight, height (only at baseline),
  * Electrocardiogram,
  * Adverse event evaluation,
  * Eastern Cooperative Oncology Group (ECOG) performance status,
  * Clinical laboratory evaluation: haematology and clinical chemistry
  * Collection of concomitant medication

SECONDARY OUTCOMES:
Immune response evaluation by treatment group as a measure of efficacy | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Katsaounis Panagiotis, MD, PhD, Principal Investigator — Iaso General Hospital, Athens
Locations (3):
- Greece (3):
  - 251 General Airforce Hospital, Athens
  - Iaso General Hospital, Athens
  - University General Hospital of Heraklion, Heraklion, Crete